CLINICAL TRIAL: NCT03027791
Title: Sodium Healthy Living Project
Acronym: SoHELP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Hearst Foundations (Unknown)
Responsible Party: Principal Investigator, Bernice Coleman, PhD, ACNP, Nurse Research Scientist, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00046886
Record Dates: First submitted 2016-12-23; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension
Keywords: Biosensors; Virtual Reality; Dietary Sodium
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Parishoners at HUMC (Experimental): African-American adults aged 18-85 who attend services at Holman United Methodist Church will be exposed to Group Sessions for 12 weeks and Virtual Reality for 6 weeks.
  Interventions: Behavioral: Virtual Reality; Behavioral: Group Sessions

INTERVENTIONS:
Behavioral: Virtual Reality — Participation in Virtual Reality experiences focused on a) education about the effects of high sodium foods on coronary arteries, blood pressure, the kidneys, and the cerebral vasculature, and b) stress management.
Behavioral: Group Sessions — 12 weekly group sessions that will provide education on topics related to hypertension, dietary sodium, physical activity and stress.

SUMMARY:
Subjects will participate in a 12-week church-based intervention with five separate components: 1) participation in weekly group sessions; 2) daily use of Fitbit activity tracker; 3) daily, twice a day blood pressure monitoring; 4) daily online food tracking; and 5) daily use of VR at home (starting at week 6). Participants will also receive phone contacts from nurse coaches (twice a week during the first 4 weeks, then once a week for the remaining 8 weeks), who will answer questions and provide support.

DETAILED DESCRIPTION:
Group sessions will be held weekly for a total of 12 sessions, with each session lasting approximately 90 minutes. Given that this is a church-based study, all group sessions will begin with a prayer, and spiritual messages will be woven into the study educational materials.

Study subjects will be asked to wear a Fitbit Flex 2 activity tracker during the 12 weeks of study participation during their waking and sleeping hours. A brief training on how to operate the Fitbit will occur during the first study session, and participants will be provided with the contact information of nurse coaches for troubleshooting purposes. Participants will have the option of keeping the Fitbit Flex 2 for their personal use after the study is complete.

Participants will receive a blood pressure cuff and will be asked to record their blood pressure measurements twice a day (upon awakening and before bed) during the 12 weeks of study participation. A brief training on how to correctly take and record blood pressure measurements will take place during the first study session, and participants will be provided with the contact information of nurse coaches for troubleshooting purposes. Participants will have the option of keeping the blood pressure monitor for their personal use after the study is complete.

During the first study session, participants will be introduced to a website in which they will be asked to log all meals daily during the 12 weeks of study participation. Instructions on how to use this website will be provided during the first study session, and participants will be provided with the contact information of nurse coaches for troubleshooting purposes.

Beginning at week 6, the VR component of the intervention will be introduced. Participants will be provided with Homido Mini Virtual Reality goggles, and they will be given instructions on how to operate the VR technology using their own phones. Participants will be asked to download a VR application to their personal phones, which will only be available for participants in the research study. The research team will help participants manually download the app into their phones. Participants will be asked to use the VR daily, and to keep a daily log of which experiences they used on each day and for how long. Participants will have the option of keeping the VR goggles for their personal use after the study is complete.

Phone contacts will be initiated by nurse coaches based on time preferences expressed by participants. These contacts will provide opportunities for participants to share their blood pressure measurements, ask questions and discuss their progress and challenges. During the first 4 weeks of the pilot, these contacts will occur twice a week, and then weekly for the remaining of the pilot. The nurse coaches will provide their contact information in case that participants desire to contact them with questions at other times.

To identify study participants, the Pastor of Holman Methodist Church will make an announcement about the study during his weekly service and direct interested people to members of the research team for more information. Additionally, study flyers with contact information for the research team will be posted throughout the church.

ELIGIBILITY:
Inclusion Criteria:

1. Parishioners or attendee of Holman Church who volunteer to participate
2. Smartphone with internet access
3. No physical disability that would inhibit full range of motion
4. Age between 18 and 85 years
5. Women who are not pregnant
6. Able to provide informed consent

Exclusion Criteria:

1. Owner of cellular or mobile phone without internet access
2. Physical ailment(s) that would inhibit full range of motion
3. Age less than 18 years or greater than 85 years
4. Pregnant women
5. Current diagnosis of epilepsy, dementia, or other neurological disease that may prevent use of VR hardware and software via self-report
6. Sensitivity to flashing light or motion
7. Recent stroke via self-report
8. Injury to the eyes or face that prevents comfortable use of VR hardware or software, or safe use of the hardware (e.g., open sores, wounds, or skin rash on face)
9. Unable to place fitbit device on wrist
10. Unable to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Daily, up to 12 weeks
  Twice daily blood pressure measurements

SECONDARY OUTCOMES:
Physical activity | Daily, up to 12 weeks
  Minutes active in a day as calculated by Fitbit Flex 2.
Dietary sodium | Daily, up to 12 weeks
  Self-reported amount of dietary sodium in diet.
Virtual Reality use | 6 weeks
  Self-reported at-home virtual reality use.
Participant satisfaction | 12 weeks
  Self-reported satisfaction with study participation.

CONTACTS AND LOCATIONS:
Overall Officials: Bernice Coleman, PhD, ACNP, Principal Investigator — Cedars-Sinai Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown DL, Conley KM, Sanchez BN, Resnicow K, Cowdery JE, Sais E, Murphy J, Skolarus LE, Lisabeth LD, Morgenstern LB. A Multicomponent Behavioral Intervention to Reduce Stroke Risk Factor Behaviors: The Stroke Health and Risk Education Cluster-Randomized Controlled Trial. Stroke. 2015 Oct;46(10):2861-7. doi: 10.1161/STROKEAHA.115.010678. Epub 2015 Sep 15. PMID 26374480
- [Background] Schoenthaler A, Lancaster K, Midberry S, Nulty M, Ige E, Palfrey A, Kumar N, Ogedegbe G. The FAITH Trial: Baseline Characteristics of a Church-based Trial to Improve Blood Pressure Control in Blacks. Ethn Dis. 2015 Aug 7;25(3):337-44. doi: 10.18865/ed.25.3.337. PMID 26674992
- [Background] Appel LJ, Champagne CM, Harsha DW, Cooper LS, Obarzanek E, Elmer PJ, Stevens VJ, Vollmer WM, Lin PH, Svetkey LP, Stedman SW, Young DR; Writing Group of the PREMIER Collaborative Research Group. Effects of comprehensive lifestyle modification on blood pressure control: main results of the PREMIER clinical trial. JAMA. 2003 Apr 23-30;289(16):2083-93. doi: 10.1001/jama.289.16.2083. PMID 12709466
- [Background] Yeary KH, Cornell CE, Prewitt E, Bursac Z, Tilford JM, Turner J, Eddings K, Love S, Whittington E, Harris K. The WORD (Wholeness, Oneness, Righteousness, Deliverance): design of a randomized controlled trial testing the effectiveness of an evidence-based weight loss and maintenance intervention translated for a faith-based, rural, African American population using a community-based participatory approach. Contemp Clin Trials. 2015 Jan;40:63-73. doi: 10.1016/j.cct.2014.11.009. Epub 2014 Nov 15. PMID 25461496
- [Background] Lancaster KJ, Schoenthaler AM, Midberry SA, Watts SO, Nulty MR, Cole HV, Ige E, Chaplin W, Ogedegbe G. Rationale and design of Faith-based Approaches in the Treatment of Hypertension (FAITH), a lifestyle intervention targeting blood pressure control among black church members. Am Heart J. 2014 Mar;167(3):301-7. doi: 10.1016/j.ahj.2013.10.026. Epub 2013 Nov 6. PMID 24576512
- [Background] Kumanyika SK, Shults J, Fassbender J, Whitt MC, Brake V, Kallan MJ, Iqbal N, Bowman MA. Outpatient weight management in African-Americans: the Healthy Eating and Lifestyle Program (HELP) study. Prev Med. 2005 Aug;41(2):488-502. doi: 10.1016/j.ypmed.2004.09.049. PMID 15917045
- [Background] Resnicow K, Jackson A, Wang T, De AK, McCarty F, Dudley WN, Baranowski T. A motivational interviewing intervention to increase fruit and vegetable intake through Black churches: results of the Eat for Life trial. Am J Public Health. 2001 Oct;91(10):1686-93. doi: 10.2105/ajph.91.10.1686. PMID 11574336
- [Background] Walker J, Ainsworth B, Hooker S, Keller C, Fleury J, Chisum J, Swan P. Optimal Health (Spirit, Mind, and Body): A Feasibility Study Promoting Well-Being for Health Behavior Change. J Relig Health. 2015 Oct;54(5):1681-98. doi: 10.1007/s10943-014-9890-7. PMID 24985320
- [Background] Schwingel A, Galvez P. Divine Interventions: Faith-Based Approaches to Health Promotion Programs for Latinos. J Relig Health. 2016 Dec;55(6):1891-906. doi: 10.1007/s10943-015-0156-9. PMID 26541338
- [Background] Lancaster KJ, Carter-Edwards L, Grilo S, Shen C, Schoenthaler AM. Obesity interventions in African American faith-based organizations: a systematic review. Obes Rev. 2014 Oct;15 Suppl 4:159-76. doi: 10.1111/obr.12207. PMID 25196412
- [Background] Horowitz CR, Goldfinger JZ, Muller SE, Pulichino RS, Vance TL, Arniella G, Lancaster KJ. A model for using community-based participatory research to address the diabetes epidemic in East Harlem. Mt Sinai J Med. 2008 Jan-Feb;75(1):13-21. doi: 10.1002/msj.20017. PMID 18306238
- [Background] Malloy KM, Milling LS. The effectiveness of virtual reality distraction for pain reduction: a systematic review. Clin Psychol Rev. 2010 Dec;30(8):1011-8. doi: 10.1016/j.cpr.2010.07.001. Epub 2010 Jul 13. PMID 20691523
- [Background] Hua Y, Qiu R, Yao WY, Zhang Q, Chen XL. The Effect of Virtual Reality Distraction on Pain Relief During Dressing Changes in Children with Chronic Wounds on Lower Limbs. Pain Manag Nurs. 2015 Oct;16(5):685-91. doi: 10.1016/j.pmn.2015.03.001. Epub 2015 May 9. PMID 25972074
- [Background] Chen X, Wang Y. Tracking of blood pressure from childhood to adulthood: a systematic review and meta-regression analysis. Circulation. 2008 Jun 24;117(25):3171-80. doi: 10.1161/CIRCULATIONAHA.107.730366. Epub 2008 Jun 16. PMID 18559702
- [Background] Atkinson NL. Developing a questionnaire to measure perceived attributes of eHealth innovations. Am J Health Behav. 2007 Nov-Dec;31(6):612-21. doi: 10.5555/ajhb.2007.31.6.612. PMID 17691874
- See also: Tables of Summary Health Statistics for U.S. Adults: 2015 National Health Interview Survey. National Center for Health Statistics — http://www.cdc.gov/nchs/nhis/SHS/tables.htm.
- See also: Building Strong Partnerships for Progress, 2012. U.S. Department of Health and Human Services — https://millionhearts.hhs.gov/files/MH_YearinReview_2012.pdf